CLINICAL TRIAL: NCT01507103
Title: A Multi-center, Randomized, Open-label, Mechanism of Action Trial on the Biological Effects of the Therapeutic Cancer Vaccine Stimuvax® (L-BLP25) in Rectal Cancer Subjects Undergoing Neoadjuvant Chemoradiotherapy
Brief Title: Tecemotide (L-BLP25) in Rectal Cancer
Acronym: SPRINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 63325-013; 2011-000847-25 (EudraCT Number)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Rectal Cancer
Keywords: Tecemotide (L-BLP25); Cyclophosphamide (CPA); Mode of action; Neoplasms; Neoplasms by Site; Carcinomas; Antineoplastic Agents; Neoadjuvant; Radiotherapy Pharmacologic Actions; Immunosuppressive Agents; Immunologic Function; Therapeutic Uses; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms; Neoplasms by Site; Carcinoma | interventions — L-BLP25; Cyclophosphamide; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chemoradiotherapy+tecemotide (L-BLP25)+CPA (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Drug: cyclophosphamide (CPA); Other: Chemoradiotherapy
- Chemoradiotherapy+tecemotide (L-BLP25) (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Other: Chemoradiotherapy
- Chemoradiotherapy (Active Comparator)
  Interventions: Other: Chemoradiotherapy

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) — Subjects will receive 8 consecutive weekly subcutaneous vaccinations with 806 microgram (mcg) of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8, which will be administered concomitantly with the chemoradiotherapy, followed by a 9th subcutaneous injection 7 to 11 days prior to surgery.
  Other Names: EMD531444
  Arms: Chemoradiotherapy+tecemotide (L-BLP25); Chemoradiotherapy+tecemotide (L-BLP25)+CPA
Drug: cyclophosphamide (CPA) — A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of CPA will be given 3 days before the first tecemotide (L-BLP25) administration.
  Other Names: L01AA01; Endoxana
  Arms: Chemoradiotherapy+tecemotide (L-BLP25)+CPA
Other: Chemoradiotherapy — Radiotherapy of 45-52 grays (Gy) will be applied 5 times per week, over a minimum period of 5 weeks. Capecitabine at a dose of 825 mg/m^2, twice daily or equivalent dose of 5-fluorouracil (5-FU) will be given orally, starting at the first day of radiotherapy and given 5 to 7 days per week during the time of radiotherapy.

SUMMARY:
The objective of this mechanistic study is to determine the impact of tecemotide (L-BLP25) administration on the mucinous glycoprotein 1 - (MUC1) specific immune response in subjects with newly diagnosed rectal cancer who are eligible for neoadjuvant therapy.

Tecemotide (L-BLP25) is designed to induce an immune response that may lead to immune rejection of tumor tissues that aberrantly express MUC1 antigen. MUC1 is highly expressed in all colorectal cancers and since the adaptive immune system plays a role in the prognosis of rectal cancer, it is reasonable to speculate that tecemotide (L-BLP25) administration might boost the tumor-specific immune response and increase the number of tumor-infiltrating lymphocytes (TILs).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with histologically documented resectable rectal adenocarcinoma in Stage 2-4
2. Availability of tumor biopsy sufficient for immunological analysis
3. Indication to receive neoadjuvant concomitant chemoradiotherapy consisting of a radiation dose of 45-52 Gy and capecitabine 825 mg/m^2 orally twice daily. The use of an equivalent schedule based on 5-FU is acceptable
4. Magnetic resonance imaging small pelvis / computed tomography thorax/abdomen (or X-ray thorax) to document absence of metastatic disease. Imaging must not be older than 6 weeks prior to randomization
5. Eastern Cooperative Oncology Group performance status of 0 or 1
6. Written informed consent
7. Greater than or equal to (>=) 18 years of age

Exclusion Criteria:

1. Previous chemotherapy and/or previous radiotherapy of the pelvic region
2. Relapsing disease
3. Previous vaccination with any MUC1 vaccine and other therapeutic cancer vaccines
4. Previous organ transplantation (bone marrow or solid organs)
5. Subjects with metastatic disease (except for solitary, resectable liver or lung metastases)
6. Inadequate hematological function (that is, platelet count less than 140*10^9 per liter [/L], or white blood cell less than 2.5*10^9/L, or hemoglobin less than 90 gram per liter). Clinically significant hepatic dysfunction (that is alanine aminotransferase greater than 2.5*upper limit of normal [ULN], or aspartate aminotransferase greater than 2.5*ULN, or bilirubin greater than 1.5*ULN). Inadequate renal function (that is serum creatinine greater than 1.5*ULN)
7. Autoimmune diseases
8. Recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have hereditary or congenital immunodeficiencies
9. Clinically significant cardiac disease, for example, New York Heart Association Classes III-IV; uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction in the previous 6 months as confirmed by medical history and an electrocardiogram
10. Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Guenther, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- NKI (Nederlands Kanker Instituut), Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): Feb 2012/Dec 2013. Study completion date: Jun 2014.
Pre-assignment Details: Enrolled: 140 screened for eligibility; 16 excluded (mainly due to non-fulfillment of inclusion or exclusion criteria), 124 subjects randomized.
Groups:
- Chemoradiotherapy+Tecemotide (L-BLP25)+CPA: Single dose of cyclophosphamide (300 mg/m^2 to a maximum of 600 mg) was administered intravenously, 3 days prior to the start of vaccination, followed by weekly subcutaneous vaccinations with tecemotide (L-BLP25) (actual delivered dose was 806 mcg) administered concomitantly with chemotherapy for 8 weeks, followed by a 9th subcutaneous vaccination 7 to 11 days prior to surgery.
- Chemoradiotherapy+Tecemotide (L-BLP25): Weekly subcutaneous vaccinations with tecemotide (L-BLP25) (actual delivered dose was 806 mcg) administered concomitantly with chemotherapy for 8 weeks, followed by a 9th subcutaneous vaccination 7 to 11 days prior to surgery.
- Chemoradiotherapy: Radiotherapy of 45-52 Gy will be applied 5 times per week, over a minimum period of 5 weeks. Capecitabine at a dose of 825 mg/m^2, twice daily or equivalent dose of 5-FU will be given orally, starting at the first day of radiotherapy and given 5 to 7 days per week during the time of radiotherapy.
Period: Overall Study
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+CPA | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Started | 41 | 41 | 42
Completed | 41 | 41 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least one dose of study treatment (tecemotide [L-BLP25] or CPA).
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+CPA | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy | Total
Number analyzed (Participants) | 39 | 41 | 42 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.74) | 62.2 (10.12) | 60.3 (8.77) | 61.3 (9.84)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 14 | 10 | 33
  Male | 30 | 27 | 32 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tumor Immune Response Evaluated by Immunohistochemical (IHC) Analysis of Tumor Infiltrating Lymphocytes (TILs) at Week 14 (Post-surgery)
Description: Tumor biopsy samples were collected prior to baseline and after the surgery. The TILs were evaluated in 3 of the most abundant high-power fields (x40) per sample and the mean value considered (after excluding the lowest and the highest value). The tumor immune response was calculated as number of TILs divided by 100 tumor cells.
Time Frame: Baseline and Week 14 (post-surgery)
Population: Immunomonitoring analysis set included all subjects for whom at least the baseline ELISpot blood and tumor sample, tumor sample at surgery and pre-surgery ELISpot blood drawing are available and whose tumor biopsy at baseline is MUC1-positive. Within the data table, n=number of subjects analyzed for each category.
Measure: Mean (Standard Deviation); unit: TILs per 100 tumor cells
Groups:
- Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide: Single dose of cyclophosphamide (300 mg/m^2 to a maximum of 600 mg) was administered intravenously, 3 days prior to the start of vaccination, followed by weekly subcutaneous vaccinations with tecemotide (L-BLP25) (actual delivered dose was 806 mcg) administered concomitantly with chemotherapy for 8 weeks, followed by a 9th subcutaneous vaccination 7 to 11 days prior to surgery.
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Number analyzed (Participants) | 27 | 33 | 30
TILs per 100 tumor cells
  CD8+ (n=23, 27, 26) | 0.609 (5.4241) | 0.543 (4.5009) | 1.538 (3.9509)
  CD8+/GrB+ (n=23, 27, 26) | 0.565 (3.1646) | 0.216 (2.4187) | 0.936 (2.7649)
Statistical Analysis 1: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy; Category: CD8+ The difference between baseline and surgical tumor samples was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm C) based on an analysis of covariance (ANCOVA) model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value as covariate. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.794, type III SS F-test — Arm effect; Effect estimate = -0.04, 95% CI 2-sided [-0.72 to 0.65]
Statistical Analysis 2: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25) vs Chemoradiotherapy; Category: CD8+ The difference between baseline and surgical tumor samples was analysed and compared across the 3 treatment arms (effect estimate for Arm B vs Arm C) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value as covariate. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.794, type III SS F-test — Arm effect; Effect estimate = -0.20, 95% CI 2-sided [-0.82 to 0.43]
Statistical Analysis 3: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy+Tecemotide (L-BLP25); Category: CD8+ The difference between baseline and surgical tumor samples was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm B) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value as covariate. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.794, type III SS F-test — Arm effect; Effect estimate = 0.16, 95% CI 2-sided [-0.49 to 0.82]
Statistical Analysis 4: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy; Category: CD8+/GrB+ The difference between baseline and surgical tumor samples was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm C) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value as covariate. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.654, type III SS F-test — Arm effect; Effect estimate = 0.02, 95% CI 2-sided [-0.52 to 0.57]
Statistical Analysis 5: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25) vs Chemoradiotherapy; Category: CD8+/GrB+ The difference between baseline and surgical tumor samples was analysed and compared across the 3 treatment arms (effect estimate for Arm B vs Arm C) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value as covariate. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.654, type III SS F-test — Arm effect; Effect estimate = -0.19, 95% CI 2-sided [-0.69 to 0.31]
Statistical Analysis 6: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy+Tecemotide (L-BLP25); Category: CD8+/GrB+ The difference between baseline and surgical tumor samples was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm B) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value as covariate. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.654, type III SS F-test — Arm effect; Effect estimate = 0.21, 95% CI 2-sided [-0.31 to 0.74]

2. Primary Outcome: Immunological Response to Treatment in Relation to Microsatellite Instability (MSI) Status: Number of Subjects Per MSI Category
Description: A potential association between MSI status (present or absent) and the primary endpoints (difference from baseline to surgery in CD8+ and CD8+/GrB+ T cell infiltration) was evaluated. Determination of mismatch repair protein (MRP)-expression (hMLH1, hMSH2, hMSH6 and hPMS2) was performed for the detection of the MSI-H-phenotype by IHC and/or on tumor deoxyribonucleic acid (DNA) sample using 5 microsatellite markers (BAT-25, BAT-26, NR-21, NR-24 and MONO-27).
Time Frame: 18 weeks
Population: Immunomonitoring analysis set included all subjects for whom at least the baseline ELISpot blood and tumor sample, tumor sample at surgery and pre-surgery ELISpot blood drawing are available and whose tumor biopsy at baseline is MUC1-positive.
Measure: Number; unit: subjects
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Number analyzed (Participants) | 27 | 33 | 30
subjects
  No | 25 | 32 | 30
  Yes | 2 | 1 | 0
Statistical Analysis 1: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy; Category: CD8+ The difference in T cell infiltration from baseline to surgery was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm C) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value and MSI category as covariates. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.921, type III SS F-test; LS Means estimate = -0.03, 95% CI 2-sided [-0.73 to 0.67] — Difference between Means adjusted on covariates baseline value and MSI category
Statistical Analysis 2: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25) vs Chemoradiotherapy; Category: CD8+ The difference in T cell infiltration from baseline to surgery was analysed and compared across the 3 treatment arms (effect estimate for Arm B vs Arm C) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value and MSI category as covariates. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.921, type III SS F-test; LS Means estimate = -0.20, 95% CI 2-sided [-0.83 to 0.44] — Difference between Means adjusted on covariates baseline value and MSI category
Statistical Analysis 3: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy+Tecemotide (L-BLP25); Category: CD8+ The difference in T cell infiltration from baseline to surgery was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm B) based on an ANCOVA model. Difference from baseline = Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value and MSI category as covariates. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.921, type III SS F-test; LS Means estimate = 0.17, 95% CI 2-sided [-0.50 to 0.83] — Difference between Means adjusted on covariates baseline value and MSI category
Statistical Analysis 4: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy; Category:CD8+/GrB+ The difference in T cell infiltration from baseline to surgery was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm C) based on an ANCOVA model. Difference from baseline=Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value and MSI category as covariates. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.890, type III SS F-test; LS Means estimate = 0.02, 95% CI 2-sided [-0.54 to 0.58] — Difference between Means adjusted on covariates baseline value and MSI category
Statistical Analysis 5: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25) vs Chemoradiotherapy; Category:CD8+/GrB+ The difference in T cell infiltration from baseline to surgery was analysed and compared across the 3 treatment arms (effect estimate for Arm B vs Arm C) based on an ANCOVA model. Difference from baseline=Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value and MSI category as covariates. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.890, type III SS F-test; LS Means estimate = -0.19, 95% CI 2-sided [-0.70 to 0.31] — Difference between Means adjusted on covariates baseline value and MSI category
Statistical Analysis 6: Comparison: Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide vs Chemoradiotherapy+Tecemotide (L-BLP25); Category:CD8+/GrB+ The difference in T cell infiltration from baseline to surgery was analysed and compared across the 3 treatment arms (effect estimate for Arm A vs Arm B) based on an ANCOVA model. Difference from baseline=Surgery value-Baseline value. Adjustment was based on ANCOVA model with treatment arm as factor and baseline value and MSI category as covariates. No interaction included. Pairwise tests have been performed to compare Arm A with Arm C, Arm B with Arm C, and Arm A with Arm B; Test type: Superiority or Other; p = 0.890, type III SS F-test; LS Means estimate = 0.21, 95% CI 2-sided [-0.32 to 0.74] — Difference between Means adjusted on covariates baseline value and MSI category

3. Primary Outcome: Change From Baseline in Interferon (IFN)-Gamma Secretion of Mononuclear Cells in Response to MUC1 by Enzyme-linked Immunosorbent Spot (ELISpot) at Post-baseline
Description: IFN-gamma secretion of mononuclear cells in response to MUC1 was to be measured by ELISpot. The maximal post-baseline value out of Week 5, Week 11-13 (pre-surgery), and Week 16-18 (follow-up / end-of trial) was evaluated in comparison to Baseline.
Time Frame: Baseline, Week 5, Week 13 (pre-surgery), and Week 18 (end-of trial)
Population: Data were not analyzed as no acceptable ELISpot assay is available
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Peritumoral Immune Response at Week 14 (Post-surgery)
Description: Immunological changes in the tumor microenvironment were evaluated based on IHC expression of CD3+, CD4+, and Ki67+CD3+ T cells; regulatory T cells (FOXP3+) and myeloid-derived suppressor cells (CD33+CD14-); other immune cells such as NK cells (CD3-CD57+), B cells (CD20+), macrophages (CD68+), and dendritic cells (S100+). Peritumoral immune response was calculated as number of lymphoid cells at the margin of the tumor or in the tumor bed (if there is complete pathological response).
Time Frame: Baseline and Week 14 (post-surgery)
Population: The pre-specified statistical threshold for reporting of results of planned analysis for either arm or interaction effect was not met in the analysis population. Hence the data was not assessed for the outcome measure.
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Immunological Response in Peripheral Blood at Week 18 (Follow-up / end-of Trial)
Description: Immunological changes in peripheral blood were evaluated based on fluorescence analysis cell sorter phenotypic characterization of T cells (CD3+CD4+ and CD3+CD8+) and of markers of activation and proliferation (CD27, BTLA); and regulatory cells such as CD3+CD4+ (or CD8+) CD45RA+CD25+FoxP3+CD127 T cells. Immunological Response in peripheral blood was measured on a continuous scale.
Time Frame: Baseline and Week 18 (follow-up / end-of trial)
Population: Immunomonitoring analysis set included all subjects for whom at least the baseline ELISpot blood and tumor sample, tumor sample at surgery and pre-surgery ELISpot blood drawing are available and whose tumor biopsy at baseline is MUC1-positive. Within the data table, n=number of subjects analysed for each category.
Measure: Mean (Standard Deviation); unit: log2 (percentage of T cells)
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Number analyzed (Participants) | 27 | 33 | 30
log2 (percentage of T cells)
  CD3-CD56+CD16+GranzymeB+ (n=26,30,24) | -0.013 (0.1051) | -0.046 (0.1259) | -0.081 (0.2238)
  CD3-CD56+CD16+Perforin+ (n=26,30,24) | -0.050 (0.0769) | -0.033 (0.1868) | -0.088 (0.2282)
  CD3+CD4+CD27+ (n=26,30,24) | -0.181 (0.1848) | -0.135 (0.1521) | -0.099 (0.1913)
  CD3-CD56+CD16+Granzyme B+/LY (n=26,30,24) | 0.264 (0.5885) | 0.047 (1.2787) | 0.415 (0.6040)
  CD3-CD56+CD16+Perforin+/LY (n=26,30,24) | 0.226 (0.5669) | 0.058 (1.2902) | 0.411 (0.6019)
  CD3-CD56+CD16-CD107a+ (n=26,30,24) | 0.216 (1.2010) | -0.318 (1.5863) | 0.037 (1.0191)
  CD3+CD8+CD127-FoxP3-CD45RA-CD25+CTLA4+(n=27,29,24) | 0.050 (0.3933) | 0.152 (0.5386) | -0.012 (0.5202)
  CD3+CD56+CD16-Granzyme B+ (n=26,30,24) | 0.479 (1.6943) | -0.241 (0.9628) | -0.024 (0.6623)
  CD3-CD56+CD16+/LY (n=26,30,24) | 0.277 (0.5448) | 0.090 (1.2968) | 0.497 (0.6119)
  CD3-CD19+BTLA4+ (n=27,29,23) | -0.030 (0.0489) | -0.028 (0.0550) | -0.017 (0.0352)
  Lymphs Tube 2 (n=27,30,25) | -1.024 (0.4392) | -0.941 (0.6080) | -0.952 (0.4761)
  CD3+CD56+CD16+CD107a+ (n=26,30,24) | -1.216 (4.5484) | 1.966 (6.6322) | -2.752 (6.4790)
  CD3+CD4+BTLA4+ (n=26,30,24) | 0.063 (1.4413) | 0.122 (0.4833) | -0.035 (0.4117)
  Lymphs Tube 3 (n=27,30,25) | -0.994 (0.4545) | -0.920 (0.5923) | -0.936 (0.4746)
  CD3+CD56+CD16+CCR7+ (n=26,30,24) | -1.341 (4.1442) | 0.541 (6.3502) | -3.390 (5.1877)
  CD3+CD8+CD127+FoxP3-CD25-CD45RA+CTLA4-(n=27,29,24) | -0.604 (0.8102) | -1.062 (1.1436) | -0.940 (1.2678)
  Background corrected CD3+CD4+IFNg+ (n=21,27,21) | 0.058 (0.9767) | 0.544 (0.9521) | 0.359 (1.3187)
  CD3+CD56+CD16+Granzyme B+/LY (n=26,30,24) | 0.243 (0.6969) | -0.201 (1.0731) | 0.131 (0.7652)
  CD3+CD56+CD16+Perforin+/LY (n=26,30,24) | 0.240 (0.6997) | -0.177 (0.9920) | 0.101 (0.7617)
  CD3+CD4+CD127+FoxP3-CD45RA-CD25+CTLA4+(n=27,29,24) | 0.711 (1.3825) | 0.674 (1.2689) | 1.035 (1.4996)

6. Primary Outcome: Change From Baseline in IFN-gamma Secretion of Mononuclear Cells in Response to Carcinoembryonic Antigen (CEA) by ELISpot at Post-baseline
Description: IFN-gamma secretion of mononuclear cells in response to CEA was to be measured by ELISpot. The maximal post-baseline value out of Week 5, Week 11-13 (pre-surgery), and Week 16-18 (follow-up / end-of trial) was evaluated in comparison to Baseline.
Time Frame: Baseline, Week 5, Week 13 (pre-surgery), and Week 18 (end-of trial)
Population: Data were not analyzed as no acceptable ELISpot assay is available
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+Cyclophosphamide | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date of first signature of informed consent until the Follow-up/End-of-Trial visit (Week 18).
Description: TEAEs: AE's during treatment; absent pre-treatment (PT)/worsened relative to PT & onset dates occurring from first trial treatment till the Follow-up/EOT. Safety Analysis Set included all randomized subjects; received at least 1 dose of treatment (arm A:one dose of CPA, arm B:one s.c. injection of tecemotide, arm C:neo-adjuvant chemoradiotherapy).
Arm/Group | Chemoradiotherapy+Tecemotide (L-BLP25)+CPA | Chemoradiotherapy+Tecemotide (L-BLP25) | Chemoradiotherapy
Serious Adverse Events (participants affected / at risk) | 10/39 | 10/41 | 12/42
Other Adverse Events (participants affected / at risk) | 38/39 | 41/41 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiotherapy+Tecemotide (L-BLP25)+CPA (N=39) | Chemoradiotherapy+Tecemotide (L-BLP25) (N=41) | Chemoradiotherapy (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiotherapy+Tecemotide (L-BLP25)+CPA (N=39) | Chemoradiotherapy+Tecemotide (L-BLP25) (N=41) | Chemoradiotherapy (N=42)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 8 (8) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 5 (5) | 3 (3) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4) | 7 (7)
Defaecation urgency (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 18 (18) | 21 (21)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Faecal incontinence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 12 (12) | 13 (13)
Painful defaecation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 10 (10) | 14 (14) | 12 (12)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4)
Rectal tenesmus (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4) | 2 (2)
Asthenia (General disorders) | 9 (9) | 7 (7) | 6 (6)
Chills (General disorders) | 4 (4) | 2 (2) | 1 (1)
Fatigue (General disorders) | 12 (12) | 9 (9) | 12 (12)
Influenza like illness (General disorders) | 4 (4) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 11 (11) | 0 (0)
Injection site haematoma (General disorders) | 2 (2) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 4 (4) | 2 (2) | 0 (0)
Injection site nodule (General disorders) | 5 (5) | 11 (11) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 7 (7) | 7 (7) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 8 (8) | 3 (3) | 7 (7)
Radiation skin injury (Injury, poisoning and procedural complications) | 2 (2) | 9 (9) | 2 (2)
Antinuclear antibody increased (Investigations) | 4 (4) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 2 (2) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 6 (6) | 13 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2)
Dysuria (Renal and urinary disorders) | 10 (10) | 8 (8) | 5 (5)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 5 (5) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Not all efficacy data were analyzed as no acceptable ELISpot assay is available. The Sponsor decided to discontinue the development of tecemotide (L-BLP25) in September 2014

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator will inform the Sponsor in advance about any plans to publish or present data from the trial. Any publications and presentations of the results (abstracts in journals or newspapers, oral presentations, etc.), either in whole or in part, by Investigators or their representatives will require pre-submission review by the Sponsor.

The Sponsor will not suppress or veto publications, but maintains the right to delay publication in order to protect intellectual property rights.